CLINICAL TRIAL: NCT06794138
Title: The Success of Implant-borne Prostheses Following Fully-guided Static Computer-assisted Implant Surgery, a Retrospective Study.
Brief Title: The Success of Implant-borne Prostheses Following Fully-guided Static Computer-assisted Implant Surgery.
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Marton Kivovics, associate professor, Semmelweis University
Other Study IDs: SEDCD56
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Edentulism
Keywords: computer assisted implant surgery; static navigation; dental implant; overdentures; fixed partial dentures; implant placement accuracy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- static Computer Assisted Implant Placement: Patients who received implant-borne prostheses following fully guided sCAIS at the Department of Public Dental Health, Semmelweis University were included in this retrospective observational study.
  Interventions: Procedure: dental implant placement

INTERVENTIONS:
Procedure: dental implant placement — The fit of the surgical guide was checked and a flapless procedure was performed under local anesthesia. However, in cases where the width of keratinized mucosa was insufficient a limited full-thickness flap was elevated. The surgical template was fixed on the remaining dentition and mucosa using template fixation pins. Fully guided implant bed preparation was performed. Osteotomies were carried out with external cooling at a drill rotation speed of 800 rpm. Implant placement was performed using a manual torque wrench Dental implants were placed non-submerged. In cases of flap elevation, wound margins were stabilized with single interrupted sutures. Sutures were removed at 7 days postop.

SUMMARY:
This study aims to determine the success of implant-borne prostheses and the accuracy of implant placement that can be achieved using fully guided static Computer Assisted Implant Surgery (sCAIS). Additional aims included the evaluation of the stability and health of hard and soft tissues, respectively surrounding the dental implants.

DETAILED DESCRIPTION:
Surgical planning A virtual planning software is used for surgical planning. Cone beam computed tomography (CBCT) reconstruction and intraoral scans are registered. Prosthetic plans are created in the software, or the radiological template was used as one. The angulation and position of the dental implants are determined by the prosthetic plan.

Surgical guides The surgical templates are manufactured by rapid prototyping (3D printing). To guide the drills for implant bed preparation sleeves are inserted in the surgical guides.

Surgical protocol Surgical interventions are performed by a single clinician experienced in dental implant placement and static navigation. Patients rinse with 0.2% chlorhexidine solution for 1 min before surgery. The fit of the surgical guide is checked under local anesthesia. Fully guided implant bed preparation is performed. Dental implants are placed non-submerged. Sutures are removed at 7 days postop. The prosthetic stages of treatment begin after a two-month healing period.

Prosthetic procedures Implant-borne overdentures are manufactured using a hybrid (analog-digital) workflow. An open tray impression is taken using a medium body silicone impression material to capture the position of the implant platforms. An overdenture and a bar mesostructure are manufactured by the dental laboratory with a precision attachment.

Fixed partial dentures (FPD) are manufactured using either a hybrid or a digital workflow. An open tray impression is taken using a medium body silicone impression material or postoperative intraoral scans are performed with scan bodies to capture the position of the implant platforms. Screw or cement-retained porcelain fused to metal FDPs are manufactured by the dental laboratory. Pre-contacts are finished using articulating papers until balanced occlusion in cases of overdentures or lateral guidance in cases of FPDs are obtained. Patients are recalled twice per year for controls and professional dental hygiene intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received implant-borne prostheses for oral rehabilitation.
* Patients who had dental implants placed using fully guided sCAIS.

Exclusion Criteria:

* patients who had major systemic diseases as classified by the American Society of Anesthesiologists (ASA grades III-IV)
* psychiatric contraindications
* patients on medication interfering with bone metabolism, including steroid therapy and antiresorptive medication
* radiation to the head or neck region within the previous five years
* localized periapical disease, including odontogenic and nonodontogenic cysts.
* high and moderate patients with existing occlusal parafunction
* evidence of uncontrolled periodontal disease
* Alcohol Use Disorder defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5)
* recreational drug abuse
* heavy smoking (>10 cigarettes/day),
* diseases of the oral mucosa, including blisters and ulcers, red and white lesions, pigmented lesions, benign tumors of the oral cavity, and oral cancer.
* pregnancy or nursing
* poor oral hygiene as determined by a modified plaque score >30%
* unavailability for regular follow-ups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Department of Public Dental Health, Semmelweis University are included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Implant survival | 5 years
  The implant is present at the surgical site without signs of failure, mobility, and pain at the time of the follow-up
Implant success | 5 years
  According to The International Congress of Oral Implantologists (ICOI) Pisa Consensus Conference.
  Success (optimum health)
  No pain or tenderness upon function 0 mobility less than 2 mm radiographic bone loss from initial surgery No exudates in the patient's history
  II. Satisfactory survival
  No pain on function 0 mobility 2-4 mm radiographic bone loss No exudates in the patient's history
  III. Compromised survival
  May have sensitivity on function No mobility Radiographic bone loss of more than 4 mm (less than half of the length of the implant body) Probing depth of more than 7 mm May have exudates in the patient's history
  IV. Failure (clinical or absolute failure)
  Any of the following:
  Pain on function Mobility Radiographic bone loss of more than half length of the implant Uncontrolled exudate Implant no longer in mouth
Success of the implant borne prostheses | 5 years
  Prostheses with four or fewer complications (screw loosening, decementation, chipping) that could be treated chairside.

SECONDARY OUTCOMES:
Intra-operative complications | at the time of the surgery
  1. insufficient space to operate
  2. fracture of the surgical guide
  3. implant placement in an inadequate position
  4. Inadequate fit of the surgical template
  5. Inadequate stability of the surgical template
Marginal Bone Loss (MBL) | 5 years
  MBL is measured on the control panoramic radiographs using ImageJ software (National Institutes of Health, Bethesda, MD, U.S.A.) by calibrating the measurement tool with the known length of the implant. Marginal bone loss was measured as the average value of the distance from the platform of the implant to the most coronal bone-to-implant contact on the mesial and distal aspects of each implant in mm.
Biomechanical complications | 5 years
  The presence or absence of biomechanical complications of the implant-borne prostheses observed during follow-up.
  1. screw loosening
  2. screw fracture
  3. implant fracture
  4. abutment fracture
  5. fracture of the mesostructure
  6. decementation
  7. chipping of the restoration
  8. fracture of the prosthesis
  9. decreased retention reported by the patient due to the wear of the matrices
  10. loss of matrices
Implant placement accuracy (Apical Global Deviation) | 2 months
  The 3D deviation between the planned and the placed implants at the center of the implant apex in mm.
Implant placement accuracy (Coronal Global Deviation) | 2 months
  The 3D deviation between the planned and the placed implants at the center of the implant platform in mm.
Implant placement accuracy (Angular deviation) | 2 months
  Angular deviation of the implant axis between planned and clinically achieved implant positions in degrees.
Peri-implant mucositis | 5 years
  Presence of peri-implant signs of inflammation (redness, swelling, line or drop of bleeding within 30s following probing) combined with no additional bone loss following initial healing
Peri-implantitis | 5 years
  Radiographically determined vertical bone loss ≥3 mm in combination with bleeding on probing (BOP) and probing depths (PD) ≥ 6 mm were deemed to indicate peri-implantitis.

CONTACTS AND LOCATIONS:
Overall Officials: Márton Kivovics, DMD, Principal Investigator — Semmelweis University
Locations (1):
- Department of Public Dental Health, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published after de-identification.
Supporting Information: Study Protocol
Time Frame: Immediately after publication, no end date.
Access Criteria: Anyone who wishes to access the data.